CLINICAL TRIAL: NCT05086783
Title: A Multicentre, Randomized Controlled Trial to Assess Video-based Feedback for Surgical Coaching in Gynecology and Gynecologic Oncology
Brief Title: Video-based Coaching (VBC) in Gynecologic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Evan Tannenbaum, Assistant Professor, Obstetrician/Gynecologist, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 3629
Record Dates: First submitted 2021-09-28; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Education; Surgery; Gynecologic Cancer
Keywords: Surgical education; Coach; Laparoscopy; Gynecologic surgery
MeSH Terms: interventions — Sarcoglycans

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the intervention (video-based coaching plus standard surgical teaching following the master-apprentice model) or the control (standard surgical teaching following the master-apprentice model)
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, the participants and the surgical coach will not be blinded. The participants will be informed of their assignment after completing the first attempt. The staff surgeon in the operating room for each attempt will be blinded. The experienced laparoscopists who will be scoring the videos will be blinded to the group allocation and the attempt number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-based coaching (Experimental): Participants in the intervention arm will receive the standard surgical teaching while in the operating room (master-apprentice model (MAM)), plus the intervention of reviewing the recorded video with the surgical coach after performing their first attempt at laparoscopic closure of the vaginal vault.
  Interventions: Other: Video-based coaching; Other: Standard surgical teaching (master-apprentice model - (MAM))
- Standard surgical teaching (Placebo Comparator): Participants in the control arm will receive the standard surgical teaching while in the operating room (master-apprentice model-(MAM)).
  Interventions: Other: Standard surgical teaching (master-apprentice model - (MAM))

INTERVENTIONS:
Other: Video-based coaching — The coaching session will follow the Wisconsin Coaching Framework (Greenberg 2015). The surgical coaching session will last at maximum 30 minutes and will occur within 1-2 week following the procedure. The surgical coaching session will occur over Zoom. The second attempt will occur within 1 week following the coaching session.
  Arms: Video-based coaching
Other: Standard surgical teaching (master-apprentice model - (MAM)) — Standard surgical teaching that conventionally occurs in the operating room follows a master-apprentice model (MAM).

SUMMARY:
This multi-centre, randomized controlled trial aims to assess the role of video-based coaching (VBC) in residency education in gynecologic and gynecologic oncology surgery. It involves a trainee and a surgical coach, who together review a recording of the trainee performing a surgical skill or procedure and coaching is provided for skill improvement. Resident performance will be evaluated using a standardized scoring scale by two experienced surgeons before and after the intervention and compared to the control group receiving the standard surgical teaching curriculum.

DETAILED DESCRIPTION:
Achieving technical excellence is a core component of surgical training. Historically, a combination of didactic teaching, surgical simulation and the master-apprentice model (MAM) were the cornerstone of surgical education. With restrictions on resident duty hours and operating time with the COVID-19 pandemic and a shift to competency-based medical education, there is an opportunity to transform surgical education and improve educational efficiency. The purpose of this study is to assess the effect of video-based coaching (VBC) on resident skill acquisition in laparoscopic suturing of the vaginal vault at the time of laparoscopic hysterectomy.

Participants will include year 3 to 5 Obstetrics and Gynecology residents completing gynecology and gynecologic oncology rotations at the study sites. Participants will be randomized to the control (standard surgical curriculum) and intervention (standard curriculum and VBC) arms on the day of the first attempt. The effectiveness of VBC will be measured by the difference in baseline and post-intervention standardized blinded score between the intervention and control group during laparoscopic closure of the vaginal cuff.

All residents will be video recorded performing laparoscopic closure of the vaginal cuff at the time of hysterectomy using video recording built into the laparoscopic equipment in the operating rooms. Residents in the control group will receive standard surgical teaching (MAM), then they will be video-recorded performing the skill at their second attempt. Residents in the intervention group will receive the standard surgical teaching plus the intervention of reviewing the recorded video with the surgical coach at the end of the procedure (MAM plus VBC). The surgical coach will provide specific personalized feedback on performance and suggestions for improvement following the Wisconsin Coaching Framework during their coaching session. Participants will then be recorded on their subsequent attempt.

All raw video footage will be edited to include only the relevant portion of the film. This will facilitate the assessment process (i.e., the assessors will view only the relevant footage). The edited video segments for both groups on both attempts will be scored independently using the validated surgical assessment tool by two blinded, experienced gynecologic laparoscopists to evaluate surgical performance (blinded to attempt number and randomization group). The average score between both assessors will be used for statistical analysis. The effectiveness of VBC will be evaluated by comparing the difference in assessment scores between the baseline and post-intervention scores between the control and intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Postgraduate year (PGY) 3 to 5 residents in the Obstetrics and Gynaecology program at the University of Toronto
* Completing chief gynecology rotation at Mount Sinai Hospital (MSH) and Sunnybrook Health Sciences Centre (SHSC), and gynecologic oncology rotation at University Health Network (UHN) and SHSC form Sept 2021 until June 2022

Exclusion Criteria:

* Previous participation in study on another rotation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in modified-OSATS (Objective Structured Assessment of Technical Skill) score after video-based coaching intervention compared to control of standard surgical teaching | The first and second attempt will occur within a 1 month timeframe. The blinded assessors will complete the evaluation of the surgical videos for performance within 6 months of study completion.
  The modified OSATS score is a standardized rubric for assessing technical skills

SECONDARY OUTCOMES:
Participant assessment of desirability of video-based surgical coaching | Desirability will be calculated at the end of study enrolment within 1 year,
  Desirability of the intervention will be evaluated based on the proportion of eligible residents who enrol in the study (number enrolled/number eligible).
Participant assessment of usefulness of video-based surgical coaching | Questionnaire to be completed by participant within 1 month of second attempt.
  Participants in the intervention arm will complete a surgical coachee questionnaire to determine if the participants in the intervention arm found the coaching experience to be useful for developing their surgical skills.
Surgical coach assessment of feasibility of video-based surgical coaching | Questionnaire to be completed by surgical coach on day of coaching session and all questionnaires will be completed within 1 year.
  Surgical coach will complete a questionnaire immediately after the coaching activity, which will collect time for video-editing, time for coaching session and receptivity of the participant to coaching
Inter-rater reliability of the video evaluations by the blinded, experienced laparoscopists | The blinded assessors will complete the evaluation of the surgical videos for performance within 6 months of study completion.
  The intraclass correlation coefficient (ICC) between the two score for each video will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Evan Tannenbaum, MD, MSc, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (3):
- Canada (3):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No